CLINICAL TRIAL: NCT04283240
Title: Pulmonary Vasodilation by Sildenafil in Acute Pulmonary Embolism
Brief Title: Sildenafil in Acute Pulmonary Embolism
Acronym: YGGDRASIL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1-10-72-282-14
Record Dates: First submitted 2020-02-07; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment was blinded by the institutional pharmacy embedding the placebo or treatment pill in a gelatinous cap
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sildenafil (Active Comparator): 50 mg sildenafil oral. One dose
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Placebo pill. One dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — 50 mg sildenafil, one dose
  Arms: Sildenafil
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To investigate if acute pulmonary vasodilation by sildenafil improves right ventricular function in patients with acute intermediate-high risk pulmonary embolism (PE).

DETAILED DESCRIPTION:
Patients with PE randomized to a single oral dose of sildenafil 50mg (n=10) or placebo (n=10) as add-on to conventional therapy. Right ventricular function evaluated immediately before and shortly after (0.5-1.5h) randomization by right heart catheterization (RHC), trans-thoracic echocardiography (TTE), and cardiac magnetic resonance (CMR). The primary efficacy endpoint was cardiac index measured by CMR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute pulmonary embolism confirmed by contrast enhanced computed tomography (CT)
* symptom duration of less than 14 days
* older than 18-80 years
* right ventricular/left ventricular ratio (RV/LV) >1 measured by trans-thoracic echocardiography (TTE, 1 cm above the atrio-ventricular valves in the four-chamber view at end-diastole).

Exclusion Criteria:

* pregnant
* cardiac arrest that required cardiopulmonary resuscitation
* a life expectancy <120 days
* systolic blood pressure <90 mmHg
* metal implants, obesity or claustrophobia that excluded the patient from cardiac magnetic resonance (CMR)
* altered mental status making the patient unable to provide informed consent
* recent use of drugs with influence on the Nitric oxide-cyclic guanosine monophosphate pathway
* known or suspected chronic thromboembolic pulmonary hypertension
* inability to perform study protocol < 72 hours after conventional PE treatment was instituted
* active bleeding after thrombolysis.

Ages: 80 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Cardiac Index | 74 (plus/minus 17) minutes after drug administration
  Cardiac Index measured by cardiac magnetic resonance imaging

OTHER OUTCOMES:
Right ventricular stroke volume | 74 (plus/minus 17) minutes after drug administration
  Evaluated by cardiac magnetic resonance imaging
Cardiac output | 74 (plus/minus 17) minutes after drug administration
  Evaluated by cardiac magnetic resonance imaging
Right ventricular end diastolic volume | 74 (plus/minus 17) minutes after drug administration
  Evaluated by cardiac magnetic resonance imaging
Right ventricular end systolic volume | 74 (plus/minus 17) minutes after drug administration
  Evaluated by cardiac magnetic resonance imaging
Right ventricular ejection fraction | 74 (plus/minus 17) minutes after drug administration
  Evaluated by cardiac magnetic resonance imaging
Mean longitudinal strain | 74 (plus/minus 17) minutes after drug administration
  Evaluated by cardiac magnetic resonance imaging
Mean pulmonary capillary wedge pressure | 32 (plus/minus 5 min) minutes after drug administration
  Evaluated by Right heart catheterization
diastolic pulmonary artery pressure | 32 (plus/minus 5 min) minutes after drug administration
  Evaluated by Right heart catheterization
systolic pulmonary artery pressure | 32 (plus/minus 5 min) minutes after drug administration
  Evaluated by Right heart catheterization
mean pulmonary artery pressure | 32 (plus/minus 5 min) minutes after drug administration
  Evaluated by Right heart catheterization
Pulmonary vascular resistance | 32 (plus/minus 5 min) minutes after drug administration
  Evaluated by Right heart catheterization
Venous oxygen saturation | 32 (plus/minus 5 min) minutes after drug administration
  Evaluated by Right heart catheterization
Right ventricular/left ventricular diameter | 84 (plus/minus 40) minutes after drug administration
  Evaluated by echocardiography
Right ventricular fractional area change | 84 (plus/minus 40) minutes after drug administration
  Evaluated by echocardiography
Tricuspid annular plane systolic excursion | 84 (plus/minus 40) minutes after drug administration
  Evaluated by echocardiography
Pulmonary artery acceleration time | 84 (plus/minus 40) minutes after drug administration
  Evaluated by echocardiography
Tricuspid regurgitant gradient | 84 (plus/minus 40) minutes after drug administration
  Evaluated by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Asger Andersen, MD,PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
By request

REFERENCES:
- [Derived] Andersen A, Waziri F, Schultz JG, Holmboe S, Becker SW, Jensen T, Sondergaard HM, Dodt KK, May O, Mortensen UM, Kim WY, Mellemkjaer S, Nielsen-Kudsk JE. Pulmonary vasodilation by sildenafil in acute intermediate-high risk pulmonary embolism: a randomized explorative trial. BMC Pulm Med. 2021 Feb 28;21(1):72. doi: 10.1186/s12890-021-01440-7. PMID 33639897